CLINICAL TRIAL: NCT05851820
Title: Prevalence and Impact of Diabetes Mellitus in Hospitalized COVID-19 Patients in a Tunisian Center: a Cross Sectional Study
Brief Title: Prevalence and Impact of Diabetes Mellitus in Hospitalized COVID-19 Patients in a Tunisian Center
Status: Completed | Type: Observational
Sponsor: Sana Rouis (Other)
Responsible Party: Sponsor-Investigator, Sana Rouis, Assistant professor in Infectious Diseases, Faculty of Medicine, Sousse
Organization: Faculty of Medicine, Sousse (Other)
Other Study IDs: SRouis
Record Dates: First submitted 2023-05-05; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Prevalence; Diabetes Mellitus; Impaction; COVID-19
Keywords: diabetes mellitus; death; complications; COVID-19; SARS-CoV2; Intensive Care Units; Tunisia
MeSH Terms: conditions — Diabetes Mellitus; COVID-19; Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic patients with COVID-19: patients hospitalized for COVID-19 and were diabetic
  Interventions: Other: comparison of outcomes/exposure
- Non-diabetic patients with COVID-19: patients hospitalized for COVID-19 and were not diabetic
  Interventions: Other: comparison of outcomes/exposure

INTERVENTIONS:
Other: comparison of outcomes/exposure — analysing if diabetes mellitus have an impact on the primary outcomes: hospital stay, admission to the ICU, death.

SUMMARY:
Objective: The objective of this study was to evaluate the prevalence and impact of diabetes mellitus on the severity and mortality of COVID-19.

Methods: Data of laboratory-confirmed hospitalized patients at the COVID-19 unit of Ibn El Jazzar University Hospital in Kairouan between September 2020 and August 2021 were analysed, in a cross-sectional study. The population was classified into two groups (COVID-19 patients with versus without diabetes). Primary outcomes were the overall length of hospital stay, the admission to the intensive care unit (ICU), and death.

DETAILED DESCRIPTION:
The outbreak of the coronavirus disease 2019 (Covid-19) has become an evolving worldwide health crisis. With the rising prevalence of diabetes mellitus has come an increasing awareness of their impacts on infectious diseases, and the risk for post-infection complications and mortality from critical infections.

Objective: The objective of this study was to evaluate the prevalence and impact of diabetes mellitus on the severity and mortality of COVID-19.

Methods: Data of laboratory-confirmed hospitalized patients at the COVID-19 unit of Ibn El Jazzar University Hospital in Kairouan between September 2020 and August 2021 were analysed, in a cross-sectional study. The population was classified into two groups (COVID-19 patients with versus without diabetes). Primary outcomes were the overall length of hospital stay, the admission to the intensive care unit (ICU), and death. Association between diabetes and death was assessed in a Cox proportional hazards model.

ELIGIBILITY:
Inclusion Criteria:

Confirmed cases indicated the patients whose real-time reverse transcriptase-polymerase chain reaction (RT-PCR) analysis results for nasal swab specimens were positive.

Exclusion Criteria:

* the investigators didn't included patients who were suspected cases, and whose the result of PCR test was negative ; Covid-19 patients admitted in other departments (Cardiology, pediatrics, obstetrics, intensive care unit, medicine, surgery department…) ; and patients with missing medical records. -

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data collection is carried out from the medical records of patients using a standardized data collection form performed by the preventive medicine department of Ibn Al Jazzar's University Hospital. A trained team of family medicine residents accomplished the data collection. The variables included the following : Socio-demographic data, underlying comorbidities, symptoms and signs at admission, routine laboratory results, complications, treatment and outcomes.
  Patients were labelled as having diabetes mellitus if they were presently treated with insulin or oral hypoglycemic agents, and based on the patient's self-report on admission
Sampling Method: Non-Probability Sample
Enrollment: 866 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Admission to Intensive Care Units | 7 days
  patients who were transferred to ICU
death | 7 days
  patients who were dead
overall length of hospital stay | 7 days
  length of hospital stay from admission to discharge (or transfer or death)

CONTACTS AND LOCATIONS:
Overall Officials: sana rouis, MD, Principal Investigator — Faculty of Medicine, Sousse
Locations (1):
- Kairouan, Kairouan, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang B, Li R, Lu Z, Huang Y. Does comorbidity increase the risk of patients with COVID-19: evidence from meta-analysis. Aging (Albany NY). 2020 Apr 8;12(7):6049-6057. doi: 10.18632/aging.103000. Epub 2020 Apr 8. PMID 32267833
- [Background] Apicella M, Campopiano MC, Mantuano M, Mazoni L, Coppelli A, Del Prato S. COVID-19 in people with diabetes: understanding the reasons for worse outcomes. Lancet Diabetes Endocrinol. 2020 Sep;8(9):782-792. doi: 10.1016/S2213-8587(20)30238-2. Epub 2020 Jul 17. PMID 32687793
- [Background] Yang JK, Feng Y, Yuan MY, Yuan SY, Fu HJ, Wu BY, Sun GZ, Yang GR, Zhang XL, Wang L, Xu X, Xu XP, Chan JC. Plasma glucose levels and diabetes are independent predictors for mortality and morbidity in patients with SARS. Diabet Med. 2006 Jun;23(6):623-8. doi: 10.1111/j.1464-5491.2006.01861.x. PMID 16759303
- [Background] Wu J, Zhang J, Sun X, Wang L, Xu Y, Zhang Y, Liu X, Dong C. Influence of diabetes mellitus on the severity and fatality of SARS-CoV-2 (COVID-19) infection. Diabetes Obes Metab. 2020 Oct;22(10):1907-1914. doi: 10.1111/dom.14105. Epub 2020 Jul 7. PMID 32496012
- [Background] Al-Salameh A, Lanoix JP, Bennis Y, Andrejak C, Brochot E, Deschasse G, Dupont H, Goeb V, Jaureguy M, Lion S, Maizel J, Moyet J, Vaysse B, Desailloud R, Ganry O, Schmit JL, Lalau JD. Characteristics and outcomes of COVID-19 in hospitalized patients with and without diabetes. Diabetes Metab Res Rev. 2021 Mar;37(3):e3388. doi: 10.1002/dmrr.3388. Epub 2020 Aug 18. PMID 32683744